CLINICAL TRIAL: NCT04690608
Title: Resistant Diabetic Macular Edema and Suprachoroidal Injection
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide in Resistant Diabetic Macular Edema, CRVO, Pseudophakic Cystoid Macular Edema and Diabetic Macular Edema Following Pars Plana Vitrectomy
Acronym: Resistant
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amin El Sayed Nawar, Lecturer Of Ophthalmology, Tanta university, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2412SS
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Retinal Edema
Keywords: macular edema
MeSH Terms: conditions — Papilledema; Macular Edema | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: cases of resistant diabetic macular edema and central retinal vein occlusion
Masking Description: code number will be given for each participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- resistant diabetic macular edema and central retinal vein occlusion (Experimental): * Prospective non randomized interventional study on 60 eyes of 40 patients with previously diagnosed macular edema secondary to type 1 or 2 diabetes mellitus will be included.
  * The study will be conducted from January 2021 to June 2021.
  * For transition to suprachoroidal injection of TAAC a diagnosis of resistant DME is required.
  Cases with recent onset central retinal vein occlusion less than 2 months duration will be included
  Interventions: Drug: Triamcinolone Acetonide 40Mg/Ml Inj,Susp_#1

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40Mg/Ml Inj,Susp_#1 — suprachoroidal injection of the drug in cases of resistant diabetic macular edema and central retinal vein occlusion
  Other Names: 30 gauge syringe with 24 gauge cannula

SUMMARY:
Prospective interventional study on 60 eyes of resistant diabetic macular edema and central retinal vein occlusion that will receive suprachoroidal injection of Triamcinolone Acetonide (SCTA).

DETAILED DESCRIPTION:
* Prospective non randomized interventional study on 60 eyes of 40 patients with previously diagnosed macular edema secondary to type 1 or 2 diabetes mellitus and 60 eyes with central retinal vein occlusion will be included.
* The study will be conducted from January 2021 to June 2021.
* For transition to suprachoroidal injection of Triamcinolone Acetone (TAAC) a diagnosis of resistant DME is required.
* Inclusion criteria:

Patients fulfilling one or more of the following criteria will be considered to have resistant diabetic macular edema (DME) after at least 3 consecutive monthly anti vascular endothelial growth factor (VEGF) injections in the previous 6 months: central macular thickness greater than 300 μm by spectral-domain optical coherence tomography (SD-OCT), reduction of retinal thickness by less than 10% of baseline retinal thickness, or suboptimal visual improvement (failure to gain at least 3 lines on the Snellen chart).

* The subjects included in the research will undergo the following tests and investigations:

  1. Visual acuity testing (uncorrected and best corrected).
  2. Intra ocular pressure (IOP) by applanation tonometry.
  3. Anterior segment examination by slit lamp
  4. Posterior segment examination by indirect ophthalmoscope and 78 D lens
  5. Spectral domain Optical coherence tomography (OCT).
  6. Ocular fundus photography and fluorescein angiography.
* Exclusion criteria will be:

  1. Previous intraocular surgery (except cataract surgery done more than 6 months before the study).
  2. Coincident retinal pathology as choroidal neovascular membrane and age related macular degeneration.
  3. Previous laser photocoagulation.
  4. Intravitreal injection of triamcinolone acetonide.
  5. Prior ocular inflammation.
  6. The presence of retinal degeneration.
  7. Patients who didnot complete 6 months of follow up

Injection technique:

Preoperative preparation:

1. Preoperative control of (Diabetes Mellitus)DM is essential before injection.
2. Informed consent was obtained according to the ethical committee after discussing extensively with each patient about the benefits, risks and possible side effects of the procedure .
3. The patient was prepared by topical fluoroquinolone eye drops (Moxifloxacin hydrochloride 0.5% Vigamox ,Alcon, USA) 4 times daily for three days before injection.

All patients were dilated before suprachoroidal injection of Triamcinolone Acetonide (SCTA) and indirect ophthalmoscope was placed at hand to examine fundus after injection.

We used 30 gauge 1cc insulin syringe. Other dispensable included 24 gauge intravenous branula. Needle was withdrawn from branula and branula was cut in such a way that only 1000um of insulin syringe was exposed from the edge of branula. 0.1 ml (4 mg ) of Triamcinolone Acetonide (TAAC) will be injected.

Post operative care:

After the injection topical antibiotic drop was applied (Moxifloxacin hydrochloride 0.5% Vigamox, Alcon, USA) and the eye was patched for several hours.

After surgery patients were instructed to administer antibiotic drop four times daily for 3 days .

* Privacy of the patients must be guaranteed ,the data acquired from the participants will stay confidential through:

  1. Putting a code number to every patient, with hiding the patient's name.
  2. Photographing faces will not be needed.
  3. The results of the research will be only used in scientific aim.
* Any unexpected risks like subconjunctival hemorrhage, syncope, vitreous hemorrhage, retinal detachment and endophthalmitis appeared during the course of the research will be cleared to the participants and the ethical committee on time.

Medical care will be carried out to complications like syncope, subconjunctival hemorrhage and surgical treatment by pars plana vitrectomy will be done in case of occurrence of vitreous hemorrhage, retinal detachment or endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling one or more of the following criteria will be considered to have resistant DME after at least 3 consecutive monthly anti VEGF injections in the previous 6 months:
* Central macular thickness greater than 300 μm by spectral-domain optical coherence tomography (SD-OCT).
* Reduction of retinal thickness by less than 10% of baseline retinal thickness.
* Suboptimal visual improvement (failure to gain at least 3 lines on the Snellen chart) and patients with recent onset central retinal vein occlusion less than 3 months.

Exclusion Criteria:

* Previous intraocular surgery (except cataract surgery done more than 6 months before the study).
* Coincident retinal pathology as choroidal neovascular membrane and age related macular degeneration.
* Previous laser photocoagulation.
* Intravitreal injection of triamcinolone acetonide.
* Prior ocular inflammation.
* The presence of retinal degeneration.
* Patients who didnot complete 6 months of follow up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of central macular thickness | 1 month
  Reduction of the central macular thickness below 300 um

SECONDARY OUTCOMES:
improved vision | 3 months
  Improvement of best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Amin E Nawar, Lecturer, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nawar AE. Efficacy of combined topical nepafenac 0.3% with suprachoroidal injection of triamcinolone acetonide using a modified custom needle in pseudopkakic cystoid macular edema. BMC Ophthalmol. 2025 Jul 3;25(1):350. doi: 10.1186/s12886-025-03972-6. PMID 40604486
- [Derived] Nawar AE. Effectiveness of Suprachoroidal Injection of Triamcinolone Acetonide in Resistant Diabetic Macular Edema Using a Modified Microneedle. Clin Ophthalmol. 2022 Nov 21;16:3821-3831. doi: 10.2147/OPTH.S391319. eCollection 2022. PMID 36438589
- [Derived] Nawar AE. Modified Microneedle for Suprachoroidal Injection of Triamcinolone Acetonide Combined with Intravitreal Injection of Ranibizumab in Branch Retinal Vein Occlusion Patients. Clin Ophthalmol. 2022 Apr 19;16:1139-1151. doi: 10.2147/OPTH.S361636. eCollection 2022. PMID 35469288